CLINICAL TRIAL: NCT04789681
Title: Single Arm Phase II Trial Using Canakinumab for the Prevention of Lung Cancer (Can-Prevent-Lung)
Brief Title: Canakinumab for the Prevention of Lung Cancer, the Can-Prevent-Lung Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-0674; NCI-2020-11724 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0674 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-12-16; First posted 2021-03-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Lung Carcinoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (canakinumab) (Experimental): Patients receive canakinumab SC on day 1. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Canakinumab; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Canakinumab — Given SC
  Other Names: ACZ885; Ilaris
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the effects of canakinumab in preventing lung cancer in patients who have high-risk pulmonary nodules. Canakinumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Giving canakinumab may prevent the development of lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether canakinumab increases regression rate of high-risk pulmonary nodules.

SECONDARY OBJECTIVES:

I. To determine whether canakinumab prolongs lung cancer-free survival. II. To determine whether canakinumab decreases the incidence of lung cancers. III. To assess the safety and tolerability of canakinumab in patients with high-risk indeterminate pulmonary nodules (IPNs).

IV. To assess quality of life by patient reported outcomes in patients treated with canakinumab.

EXPLORATORY OBJECTIVES:

I. To explore the radiographic (including radiomic features) evolution of high-risk IPNs with treatment of canakinumab and to assess their association with risks of lung cancer as well as their association with clinical benefit/toxicities in patients treated with canakinumab.

II. To explore the T-cell receptor (TCR) repertoire evolution of patients with high-risk IPNs and assess their association with risks of lung cancer as well as their association with clinical benefit/toxicities in patients treated with canakinumab.

III. To explore the evolution of serum soluble factors, such as IFN-gamma and interferon inducible factors (such as CXCL9 and CXCL10), IL-12, TNFalpha, IL-10, TGF-beta, VEGF, IL-6, IL-8, IL-17, IL-18, C-reactive protein etc.) and assess their association with risks of lung cancer as well as their association with clinical benefit/toxicities in patients treated with canakinumab.

OUTLINE:

Patients receive canakinumab subcutaneously (SC) on day 1. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed up for 30 days and at 6, 12, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant (or legally authorized representative if applicable) provides written informed consent for the trial
* Participants are eligible to be included in the study if one of the following criteria applies:

  * Patients with no history of lung cancer, who have persistent IPNs (on two computed tomography [CT] scans at least 3 months apart with no evidence of shrinkage or regression) detected by low dose computed tomography [LDCT]-guided lung cancer screening or imaging studies for other reasons (incidentalomas) with 10-30% cancer probability by Brock University cancer prediction equation as following
  * Patients with no history of lung cancer, who have persistent IPNs (on two CT scans at least 3 months apart with no evidence of shrinkage or regression) detected by LDCT-guided lung cancer screening or imaging studies for other reasons (incidentalomas) with > 30% cancer probability by Brock University cancer prediction equation as following, but biopsy showed no clear evidence of malignancy
  * Patients with history of stage I-III non-small cell lung cancer (NSCLC), who have completed treatment with curative intent, who have persistent IPNs (on two CT scans at least 3 months apart with no evidence of shrinkage or regression) with 5-30% cancer probability by Brock University cancer prediction equation as following
  * Patients with history of stage I-III NSCLC, who have completed treatment with curative intent, who have persistent IPNs (on two CT scans at least 3 months apart with no evidence of shrinkage or regression) with > 30% cancer probability by Brock University cancer prediction equation, but biopsy showed no clear evidence of malignancy
* At least 18 years of age on the day of signing informed consent
* A male participant must agree to use a contraception during the treatment period plus an additional 6months (a spermatogenesis cycle) after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 6 months after study treatments with risk of genotoxicity after the last dose of study treatment
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the start of study treatment
* Absolute neutrophil count (ANC) >= 1500/uL (collected within 10 days prior to the start of study treatment)
* Platelets >= 100 000/uL (collected within 10 days prior to the start of study treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (collected within 10 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
* Creatinine =< 1.5 x upper limit or normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (collected within 10 days prior to the start of study treatment)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (collected within 10 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x ULN (collected within 10 days prior to the start of study treatment)

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication
* Has received prior therapy with an anti-IL1beta
* Has a known additional malignancy that is progressing or has required active treatment within the past year. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has an active infection requiring systemic therapy
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through 6 months after the last dose of trial treatment
* Is receiving the following therapies during the screening and treatment phases (including retreatment for post-complete response relapse) of this trial: antineoplastic systemic chemotherapy or biological therapy, immunotherapy not specified by this protocol, chemotherapy not specified by this protocol, investigational agents other than canakinumab
* Has received live vaccines within 30 days prior to first dose of study treatment and while participating in the study. Examples of live vaccines include but are not limited to: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacillus Calmette-Guerin (BCG) and typhoid vaccine. (Note: Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (eg FluMist are live attenuated vaccines are not allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Regression of indeterminate pulmonary nodules (IPNs) | At 7 months after treatment
  Will assess complete response or partial response by modified Response Evaluation Criteria in Solid Tumors criteria.

SECONDARY OUTCOMES:
Lung cancer-free survival | Up to 24 weeks
  Will be computed using the Kaplan-Meier method.
Incidence of lung cancers | Up to 24 weeks
Incidence of adverse events | Up to 24 weeks
Quality of life questionnaires | Baseline and 24 weeks
  Assessed using The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core Questionnaire (EORTC QLQ-C30) Score ranges (1-4) 1-Not at all, 2-A little, 3-Quite a bit, 4-Very Much
Quality of life questionnaires | Baseline and 24 weeks
  Assessed using The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - the Quality of Life Lung Cancer 29 Module (EORTC QLQ-LC29).
  Score ranges (1-4) 1-Not at all, 2-A little, 3-Quite a bit, 4-Very Much

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Zhang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org